CLINICAL TRIAL: NCT05580250
Title: A Phase I, Single-Centre Study to Investigate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Doses of LY3526318, and to Investigate the Effect of LY3526318 on Metformin and Simvastatin Pharmacokinetics in Healthy Male Japanese Participants
Brief Title: A Study of LY3526318 in Healthy Male Japanese Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor made a business decision to withdraw the trial.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 18353; J2D-JE-CVAD (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Healthy
MeSH Terms: interventions — Iohexol; Simvastatin; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Part A and B are double blind and Part C is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part A: Single Dose LY3526318 (Experimental): LY3526318 administered orally in three study periods.
  Interventions: Drug: LY3526318
- Part A: Single Dose Placebo (Placebo Comparator): Placebo administered orally in three study periods.
  Interventions: Drug: Placebo
- Part B: Multiple Dose LY3526318 (Experimental): LY3526318 administered orally.
  Interventions: Drug: LY3526318
- Part B: Multiple Dose Placebo (Placebo Comparator): Placebo administered orally.
  Interventions: Drug: Placebo
- Part C: Iohexol + Simvastatin + Metformin + LY3526318 (Experimental): Iohexol administered intravenously (IV) and simvastatin, metformin, and LY3526318 administered orally.
  Interventions: Drug: LY3526318; Drug: Iohexol; Drug: Simvastatin; Drug: Metformin

INTERVENTIONS:
Drug: LY3526318 — Administered orally.
  Arms: Part A: Single Dose LY3526318; Part B: Multiple Dose LY3526318; Part C: Iohexol + Simvastatin + Metformin + LY3526318
Drug: Placebo — Administered orally.
  Arms: Part A: Single Dose Placebo; Part B: Multiple Dose Placebo
Drug: Iohexol — Administered intravenously (IV).
  Arms: Part C: Iohexol + Simvastatin + Metformin + LY3526318
Drug: Simvastatin — Administered orally.
  Arms: Part C: Iohexol + Simvastatin + Metformin + LY3526318
Drug: Metformin — Administered orally.
  Arms: Part C: Iohexol + Simvastatin + Metformin + LY3526318

SUMMARY:
This is a study of LY3526318 in healthy male Japanese. The main purposes of this study are to:

* Assess how safe and well tolerated LY3526318 is when given by mouth.
* Measure how LY3526318 affects the kidney and the liver. The study will be conducted in three parts (Part A, Part B, Part C). Participants may only enroll in one part. After screening, the study will last from one to two weeks, depending on part.

ELIGIBILITY:
Inclusion Criteria:

* Male Japanese participants who are overtly healthy as determined by medical evaluation including medical history and physical examination.
* Body weight of at least 50 kilogram (kg) and body mass index within the range 18 to 30 kilogram per square meter (kg/m2).
* Male participants must adhere to the contraceptive requirements.
* Have clinical laboratory test results within normal reference range for the population or clinical research unit (CRU), or results with acceptable deviations that are judged not clinically significant by the investigator.

Exclusion Criteria:

* Have a history or presence of medical illness including, but not limited to, any cardiovascular, hepatic, respiratory, hematological, endocrine, psychiatric or neurological disease, or convulsions that, in the judgment of the investigator, indicate a medical problem that would preclude study participation.
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study. In addition, participants with the following finding will be excluded:
* Have a history of clinically significant multiple or severe drug allergies or severe posttreatment hypersensitivity reactions.
* Show evidence of human immunodeficiency virus and/or positive human immunodeficiency virus antigens and/or antibodies, hepatitis C and/or positive hepatitis C antibody, or hepatitis B and/or positive hepatitis B surface antigen.
* Show evidence of syphilis or have a positive syphilis test.
* Have an abnormal blood pressure (supine) as determined by the investigator.
* Are unwilling to stop herbal supplements, over-the-counter, or prescription medicines, including drugs that are known inducers or inhibitors of cytochrome P450 3A4 (CYP3A4), within 14 days prior to study intervention administration and for the duration of the study. An exception is for acetaminophen at doses of less than or equal to (≤3) grams/day.
* Participated (defined as last dose of study drug) within 30 days prior to dosing in a clinical trial involving an investigational product or nonapproved use of a drug with a short half-life, or within 5 half-lives of an investigational product with a half-life longer than 6 days.
* Participants with a history of drug abuse which, in the opinion of the investigator, is clinically significant or who test positive for drugs of abuse at screening or admission.
* Are unwilling to comply with the required dietary restrictions.

Additional Exclusion Criteria of Part C:

* Have known allergies to iohexol, iodine, simvastatin, metformin, and related compounds or any components of the formulation.
* Show evidence of CYP3A5 *1 allele (CYP3A5*1/*1 or CYP3A5*1/*3).
* Confirmed creatinine clearance <90 milliliter per minute (mL/min) at the screening period assessment.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Part A and B: Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Day 12
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module.
Part C: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Metformin | Predose on Day -2 through Day 8
  PK: Cmax of metformin.
Part C: PK: Area Under the Concentration Versus Time Curve (AUC) of Metformin | Predose on Day -2 through Day 8
  PK: AUC of metformin.
Part C: PK: Total Body Clearance (CL) of Iohexol | Predose on Day -5 through Day 4
  PK: CL of Iohexol.
Part C: PK: Cmax of Simvastatin | Predose on Day -4 through Day 6
  PK: Cmax of simvastatin.
Part C: PK: AUC of Simvastatin | Predose on Day -4 through Day 6
  PK: AUC of Simvastatin.
Part C: PK: Cmax of Simvastatin Acid | Predose on Day -4 through Day 6
  PK: Cmax of Simvastatin Acid.
Part C: PK: AUC of Simvastatin Acid | Predose on Day -4 through Day 6
  PK: AUC of Simvastatin Acid.

SECONDARY OUTCOMES:
Part A, B, and C: PK: Cmax of LY3526318 | Predose on Day 1 up to Day 14
  PK: Cmax of LY3526318.
Part A, B, and C: PK: AUC of LY3526318 | Predose on Day 1 up to Day 14
  PK: AUC of LY3526318.

CONTACTS AND LOCATIONS:
Overall Officials: 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Souseikai Fukuoka Mirai Hospital, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No